CLINICAL TRIAL: NCT00632255
Title: Compliance to Long Term Imatinib Therapy in Newly Diagnosed Patients With Chronic Myeloid Leukaemia.
Brief Title: Long Term Therapy With Imatinib: Development of Late Side Effects and Compliance to Treatment
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: MADA1012
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Chronic Myeloid Leukemia; Newly Diagnosed
Keywords: Chronic Myeloid Leukemia; Long term Imatinib therapy compliance; Newly diagnosed; Late side effects
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with CML who have been treated with Imatinib (Glivec) within 6 months of diagnosis as first line therapy. Initial therapy with Hydroxyurea is permitted
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Conventional therapy with imatinib

SUMMARY:
Imatinib has revolutionised the treatment of chronic myeloid leukaemia (CML). The first clinical trials were conducted in 1998 in patients with advanced disease, and by 2002 imatinib was established as the standard therapy for all patients including those recently diagnosed. In spite of overwhelming evidence about its efficacy we still need to gain more knowledge about issues related to long term treatment with imatinib such as why some patients respond better than others, the development of side effects and the quality of life.

DETAILED DESCRIPTION:
We plan to follow prospectively a cohort of CML patients in order to study their compliance to therapy,pharmacological levels of imatinib and the prevalence of side effects. We expect to be able to correlate the actual dose received, the pharmacological levels of drug in blood, with the change in the level of residual disease (measured by Q-PCR) at various time points. We also want to gain insight into the relationship between compliance to therapy and specific side effects and between compliance and duration of treatment. We will also assess the adherence to imatinib therapy after increases in the drug dose that are part of standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CML who have been treated with imatinib (Glivec®) within 6 months of diagnosis as first line therapy. Initial therapy with hydroxyurea is permitted.

Exclusion Criteria:

* Unable to give consent.
* Unable to communicate with the medical and nursing staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CML who have been treated with imatinib (Glivec®) within 6 months of diagnosis as first line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Marin, Consultant Haematology, Study Director — Imperial College Healthcare NHS Trust
Locations (1):
- Haematology Department. Catherine Lewis Centre. Hammersmith Hospital. Du Cane Road., London, United Kingdom

REFERENCES:
- [Result] Marin D, Bazeos A, Mahon FX, Eliasson L, Milojkovic D, Bua M, Apperley JF, Szydlo R, Desai R, Kozlowski K, Paliompeis C, Latham V, Foroni L, Molimard M, Reid A, Rezvani K, de Lavallade H, Guallar C, Goldman J, Khorashad JS. Adherence is the critical factor for achieving molecular responses in patients with chronic myeloid leukemia who achieve complete cytogenetic responses on imatinib. J Clin Oncol. 2010 May 10;28(14):2381-8. doi: 10.1200/JCO.2009.26.3087. Epub 2010 Apr 12. PMID 20385986